CLINICAL TRIAL: NCT01532232
Title: Treatment of Tobacco Dependence in Breast Cancer Patients: A Randomized Trial of Varenicline (Chantix)
Brief Title: Tobacco Dependence in Breast Cancer Patients Trial of Varenicline (Chantix)
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-136
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer; Tobacco Dependence
Keywords: PLACEBO; VARENICLINE (CHANTIX); Self-reported cigarettes smokers; Smoking Cessation; 11-136
MeSH Terms: conditions — Breast Neoplasms; Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva samples

GROUPS / COHORTS (2):
- placebo: This is a randomized, double-blind, placebo-controlled trial comparing the effectiveness and tolerability of varenicline with placebo for smoking cessation in 30 tobacco dependent breast cancer patients.
  Interventions: Drug: placebo
- varenicline: This is a randomized, double-blind, placebo-controlled trial comparing the effectiveness and tolerability of varenicline with placebo for smoking cessation in 30 tobacco dependent breast cancer patients.
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: placebo — Pts will receive the standard 12-week dosing regimen consisting of 1 mg po of study drug twice daily for 11 weeks,along with smoking cessation counseling, for 11 weeks with an initial dose titration to full strength during the 1st week as follows: 0.5 mg po once daily for 3 days titrated to 0.5mg po twice daily for 4 days. 154 pills will be supplied for the 12 week tx. In order to compensate for any accidentally dropped or lost pills during the study duration, a total of 175 pills will be given to the patient. Along with smoking cessation counseling, for 11 weeks. Pts will receive their medication from the MSK Pharmacy & equivalent dosing & side effect education from our Tobacco Cessation Nurse Practitioner. Tx with the study drug will begin after the initial counseling session. Physicians & tobacco cessation nurses will be blinded regarding pts' assignment to medication or placebo tx arm. Likewise, pts will not be informed as to which medication condition they have been assigned.
  Groups: placebo
Drug: varenicline — Pts will receive the standard 12-week dosing regimen consisting of 1 mg po of study drug twice daily for 11 weeks,along with smoking cessation counseling, for 11 weeks with an initial dose titration to full strength during the 1st week as follows: 0.5 mg po once daily for 3 days titrated to 0.5mg po twice daily for 4 days. 154 pills will be supplied for the 12 week tx. In order to compensate for any accidentally dropped or lost pills during the study duration, a total of 175 pills will be given to the patient. Along with smoking cessation counseling, for 11 weeks. Pts will receive their medication from the MSK Pharmacy & equivalent dosing & side effect education from our Tobacco Cessation Nurse Practitioner. Tx with the study drug will begin after the initial counseling session. Physicians & tobacco cessation nurses will be blinded regarding pts' assignment to medication or placebo tx arm. Likewise, pts will not be informed as to which medication condition they have been assigned.
  Groups: varenicline

SUMMARY:
Breast cancer patients who smoke, are at greater risk for treatment complications. The purpose of this study is to see if the researchers can find ways to help patients who have breast cancer quit smoking. They will compare two ways to help people quit smoking. Some patients will receive varenicline, a prescription medicine also known as Chantix,®. Other patients will receive a placebo drug. A placebo is an inactive substance that contains no medicine. All patients will receive smoking cessation counseling provided by our tobacco treatment specialists. They hope that what the researchers learn from this study will help us improve our smoking cessation treatment program for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* MSK patients diagnosed with breast cancer or have a mass suspicious of breast cancer at the time of enrollment, as per clinician judgment or EMR;
* Self-reported current cigarette smoker (defined as daily smoking in the past seven days)
* Advised to quit smoking by their MSK physician and willing to receive smoking cessation counseling and treatment; as per self report
* Fluent in English

Exclusion Criteria:

* Patients less than 18 years of age because the safety and efficacy of varenicline have not yet been tested in children;
* Evidence of any known or suspected medical contraindications for use of varenicline (e.g., recent (within past two months) cardiovascular instability (including myocardial infarction or unstable angina; uncontrolled hypertension, significant neurological sequelae of cerebrovascular disease, or severe congestive heart failure (New York Heart Association class III or IV), severe chronic obstructive pulmonary disease; uncontrolled gastrointestinal, hepatic, or endocrine disease; or severe renal impairment.
* Self-reported evidence of significant psychiatric history (e.g., schizophrenia, unstable bipolar disorder, panic disorder, untreated major depression) sufficient, in the investigators' judgment, to preclude participation in the clinical trial;
* Self-reported evidence of recent substance abuse or heavy alcohol use (> 14 drinks weekly) in the last 6 months;
* Self-reported recent use (in the past 30 days) or planned use of nicotine replacement therapy (NRT) or other FDA approved cessation pharmacotherapy (bupropion);
* Pre-menopausal women who are pregnant as per EMR
* Women who are breast-feeding as per self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK breast clinic
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
effectiveness | 2 years
  To conduct a double-blind, randomized clinical trial to obtain pilot data on the the effectiveness of Intervention (varenicline and behavioral smoking cessation counseling) and Control (placebo and behavioral smoking cessation counseling) with regard to tobacco (smoking) cessation outcomes (point abstinence, continuous abstinence) in tobaccodependent breast cancer patients.

SECONDARY OUTCOMES:
examine baseline factors that are associated with poor treatment response | 2 years
  To describe the association between baseline factors (i.e., demographic, smoking history and psychosocial) and poor cessation treatment response (i.e., persistent smoking, post-surgical smoking relapse
tolerability of and adherence | 2 years
  Adherence to study medication will be assessed by summarizing the medication logs. Tolerability will be assessed by percent of patients who discontinue study medication due to side effects. Using CTCAE 4.0
rates of surgical complications | 2 years
  among tobacco dependent breast cancer patients. We will primarily use descriptive statistics to summarize the rates of surgical complications among tobacco dependent breast cancer patients, as indicated by the prevalence of surgical complications (i.e., occurrence of infection, skin flap necrosis, reconstructive flap failure, seroma, and hematoma) documented in the patient's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/